CLINICAL TRIAL: NCT07335744
Title: Construction of a Multidimensional Risk Prediction Model for Severe Early Childhood Caries Based on the "Bio-psy-social" Medical Model
Brief Title: Construction of a Multidimensional Risk Prediction Model for Severe Early Childhood Caries
Status: Not yet recruiting | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojing Li, attending doctor, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: 2026-IRB-0008-P-01
Record Dates: First submitted 2025-12-24; First posted 2026-01-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Severe Early Childhood Caries; Caries
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire survey — Parents fill out the "Children's Oral Health and Comprehensive Development Assessment Form", which includes scales such as family socioeconomic status, parental burnout in child-rearing (PBA), children's executive function (BRIEF-P), sleep habits (CSHQ), and dental fear (CFSS-DS).

SUMMARY:
This study aims to address the high prevalence and recurrence rate of severe early childhood caries (S-ECC) by breaking away from the traditional single biological factor perspective and introducing the theories of "24-hour activity behavior" and "family psychological stress". By collecting clinical and behavioral data from 1,200 preschool children and their parents, it explores the association pathways between parental burnout, children's executive function, sleep/dietary behaviors and S-ECC, and builds a high-precision risk prediction model to provide evidence-based support for the clinical development of personalized prevention strategies.

DETAILED DESCRIPTION:
Severe Early Childhood Caries (S-ECC), as a serious infectious disease that severely endangers the physical and mental health of preschool children, has now become a major public health challenge in pediatric dentistry in China. Epidemiological data show that the prevalence of caries among 3-5-year-old children in China remains high, and it is characterized by rapid disease progression, extensive tooth surface involvement, and high treatment difficulty. S-ECC not only leads to extensive tooth tissue loss in children, causing severe pain due to pulpitis and periapical inflammation, but also seriously affects children's masticatory efficiency, facial growth and development, language function, and sleep quality, and may even induce systemic diseases due to long-term chronic inflammation. Although current clinical treatment methods cover fluoride application, minimally invasive restoration, and comprehensive treatment under general anesthesia, high postoperative recurrence rates and difficult behavioral management are common problems in clinical practice. This reveals the limitations of the current "biomedical model" dominated diagnosis and treatment system, which focuses on the repair of dental lesions but neglects the deep-seated family behavioral and psychosocial roots that cause the disease and its recurrence.

Previous research on the etiology of S-ECC mainly focused on biological aspects such as cariogenic bacteria (such as Streptococcus mutans), host factors (such as saliva composition and tooth structure), and environmental factors (such as sugar intake frequency) . With the deepening of research, although some scholars have begun to pay attention to the impact of socioeconomic status (SES) on oral health, finding that parents' educational level and family income are significantly related to the caries rate, these macroscopic sociodemographic indicators are difficult to explain why there are significant differences in oral health management capabilities among families with similar socioeconomic backgrounds . The current knowledge gap lies in the lack of analysis of the family aggregation mechanism of S-ECC from the perspective of micro psychology and behavioral neuroscience. In particular, the concept of "parental burnout" proposed in the field of psychology in recent years, which refers to the emotional exhaustion and reduced parental efficacy that parents experience under long-term parenting stress, may lead to the lack or ineffectiveness of their supervision over children's oral hygiene behaviors, but this has not been fully verified in the field of dentistry . At the same time, previous studies often viewed dietary habits in isolation and ignored the "24-hour activity behavior" holistic view proposed by the World Health Organization, that is, there may be complex interactions between sleep disorders (such as mouth breathing, night waking), sedentary behavior (excessive screen time), and unhealthy diet, which together form a risk loop for S-ECC. In addition, the cognitive traits of preschool children themselves, such as deficits in inhibitory control in executive function, may lead to poor cooperation in tooth brushing and poor control of dietary impulses, and the impact of this neuro-psychological characteristic on the susceptibility to S-ECC is also a blind spot in current research.

Given the above background and research status, it is particularly urgent and important to conduct multi-dimensional risk factor research on S-ECC in preschool children based on the "biopsychosocial" medical model. This study aims to break through the framework of traditional etiological research, and on the basis of collecting objective clinical indicators such as the dmft index and plaque index, introduce psychological and behavioral science assessment tools to systematically explore the deep association pathways between parental burnout, children's executive function deficits, and unhealthy lifestyles (sleep, screen time) and the onset of S-ECC. This study not only helps to fill the current knowledge gap regarding the psychosocial pathogenesis of S-ECC and explain the phenomenon that "high-knowledge families" may still have a high risk of caries, but also has important clinical translation significance. By constructing a multi-dimensional risk prediction model of S-ECC that incorporates psychological and behavioral characteristics, clinicians can identify families with "high-risk psychological and behavioral characteristics" at an early stage, thereby moving the intervention point forward and achieving a shift from merely "tooth treatment" to "overall oral health management of the family". This provides a solid evidence-based medical basis for formulating precise personalized prevention strategies and reducing the recurrence rate of S-ECC.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 3-6 years old (36 months ≤ months < 72 months);
* Good overall health condition (ASA classification I-II);
* Parents have given informed consent and are willing to participate in this study.

Exclusion Criteria:

* Suffering from severe systemic diseases (such as congenital heart disease, blood disorders, immune deficiencies, etc.);
* Having congenital craniofacial deformities (such as cleft lip and palate, facial clefts, etc.);
* Undergoing orthodontic treatment for the mouth;
* Having a history of long-term use of drugs that affect saliva secretion;
* Refusing to undergo oral clinical examination or unable to cooperate.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who visited the oral department of the Children's Hospital affiliated to Zhejiang University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
number of carious teeth at the baseline | at the baseline
  The number of the carious teeth includes the treated or untreated carious teeth.
number of carious teeth at 6 months | at 6 months after enrollment
  The number of carious includes treated or untreated carious teeth.
number of carious teeth at 1 year | at 1 year after enrollment
  the number of carious teeth includes treated or untreated carious teeth.

IPD SHARING:
Plan to Share IPD: No